CLINICAL TRIAL: NCT05356650
Title: Comparative Effects of Mulligan's Mobilization and Proprioceptive Neuromuscular Facilitation Technique on Pain and Disability in Patients With Sacroiliac Joint Dysfunction: A Randomised Controlled Trail
Brief Title: Mulligan's Mobilization and Proprioceptive Neuromuscular Facilitation Technique in Sacroiliac Joint Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0109 Aisha
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: SACROILIAC JOINT DYSFUNCTION
Keywords: Mulligan Mobilization; Proprioceptive Neuromuscular Facilitation; Contract Relax; Sacroiliac joint Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilization (Experimental): Treatment will be given with frequency of 3 sets with 10 repetitions on sacroiliac joint 3 times a week for 6 weeks
  Interventions: Other: Mulligan Mobilization
- PNF Technique (Experimental): Three sets of stretching of each muscle will be performed for each position with the frequency of 3 times a week for 6 weeks.
  Interventions: Other: PNF

INTERVENTIONS:
Other: Mulligan Mobilization — The patient will be in a prone position. With one hand, the physiotherapist will fix the sacrum and place the fingers of her other hand under the anterior superior iliac spine. The therapist then pull the ilium on the sacrum and will instruct the patient to do press-ups. Treatment will be given with frequency of 3 sets with 10 repetitions on sacroiliac joint 3 times a week for 6 weeks
  Arms: Mulligan Mobilization
Other: PNF — PNF stretching will be performed using contract-relax techniques of agonists in supine, prone and side-lying. Contract-relax will be applied with a 6-second contraction with 80% force of the maximal isometric contraction on the muscles (iliopsoas, hamstrings and gluteal muscles) and will be followed by a 15-second passive static stretching in the opposite direction of that muscles. Three sets of stretching of each muscle will be performed for each position with the frequency of 3 times a week for 6 weeks.
  Patient will be in supine, prone, side lying. Both groups will receive a baseline treatment (Moist Heat Pack for 10 minutes and 10 minutes of Ultrasound (0.75 MHz, continuous wave)
  Arms: PNF Technique

SUMMARY:
This study will aim to compare the effects of mulligan mobilization and PNF on pain and disability with patients of SIJ dysfunction and will be helpful for clinical physiotherapist to choose more effective treatment protocol for patients as there are fewer researches on comparison of these techniques.

DETAILED DESCRIPTION:
The sacroiliac joint dysfunction syndrome (SIJDS) is an ongoing controversial issue and an important source of low back pain (LBP). It has been emphasized in many studies that the pathologies of sacroiliac joint (SIJ) are a source of pain in the lumbar spine and hip region. The prevalence of SIJDS in patients with chronic mechanical LBP is between 15 and 30% SIJD is a condition in which pain arises from the sacroiliac joint and is caused by the abnormal movement of ilium around the sacrum and abnormal function of the SIJ structures, like ligaments, muscles, capsules. The prevalence of SIJP has been stated to be up to 75% in LBP patients.

Physiotherapy techniques are used to correct SIJ mal-alignment manually by restoring the normal function and balance of lumbar and pelvic muscles and ligaments. Mulligan described the positional fault theory in which articular mal-alignment leads to altered kinematics and eventual dysfunction(2). Proprioceptive neuromuscular facilitation (PNF) is a form of flexibility exercises used to resolve muscle shortening and strain.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 35 years

  * Both genders
  * Subjects with positive provocation test ( Faber's test\Patricks test, Gaenslen test, distraction test, compression test, sacral thrust test)
  * Subjects with positive innominate test ( Stork Test\Gillet Test)
  * Subjects who agree to fill the informed consent

Exclusion Criteria:

* Pregnant women

  * Presence of neurological signs
  * Patient with ankylosis spondylosis.
  * Patient has been diagnosed by disease other than SIJ dysfunction
  * Patients having any congenital posture problem or previous surgery
  * SLR less than 45 degree
  * Patient having any mental problem or reduced cognitive ability

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating scale | 3 months
  The most common validated tool for assessment of pain in clinical tests is the numeric pain rating score (NPRS), a 10-point scale where 0 indicates no pain and 10 indicates severe pain
Modified Oswestry Disability Questionnaire | 3 months
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The questionnaire consists of 10 items addressing different aspects of function. Each item is scored from 0 to 5, with higher values representing greater disability. The total score is multiplied by 2 and expressed as a percentage

CONTACTS AND LOCATIONS:
Overall Officials: Nosheen Manzoor, Principal Investigator — Riphah International University
Locations (1):
- Govt. Hospital DHQ, Jhang, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No